CLINICAL TRIAL: NCT02675855
Title: A Multicenter, Randomized, Single-Blind Study Comparing the Efficacy of GrafixPRIME® to Active Comparator for the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: GrafixPRIME® for the Treatment of Chronic Diabetic Foot Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Osiris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protocol 350
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Foot Ulcer, Diabetic
Keywords: Grafix
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GrafixPRIME® (Experimental): GrafixPRIME® is cryopreserved human placental membrane Patients will be fitted with off-loading devices
  Interventions: Other: GrafixPRIME®; Device: Off-loading (walking boot)
- Active Comparator (Active Comparator): Wound cover, Dressing Application Patients will be fitted with off-loading devices
  Interventions: Procedure: Dressing Application; Device: Off-loading (walking boot)

INTERVENTIONS:
Other: GrafixPRIME® — Human tissue, Wound cover, Application of a non-adherent dressing, a moisture retentive dressing, and a secondary dressing.
  Arms: GrafixPRIME®
Procedure: Dressing Application — Wound cover, Application of a non-adherent dressing, a moisture retentive dressing, and a secondary dressing.
  Arms: Active Comparator
Device: Off-loading (walking boot) — Patients will be fitted for an off-loading device (walking boot) and agree to comply with use of the device during the course of the study

SUMMARY:
The objective of the study is to compare the efficacy of weekly GrafixPRIME® administration to an Active Comparator in patients with chronic DFUs in a randomized, single-blind study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 Diabetes
* Chronic ulcer (present for ≥4 weeks, but not more than 52 weeks)
* Index ulcer located below the malleoli on the plantar or dorsal surface of the foot
* Index ulcer extends into the dermis or subcutaneous tissue without evidence of exposed muscle, tendon, bone or joint capsule
* Adequate circulation to the foot (documented by ABI or TBI)

Exclusion Criteria:

* Gangrene present on affected foot
* Index ulcer is over a Charcot deformity
* Patient is receiving dialysis
* Patient has 2 or more previous amputations
* Patient has HbA1c >12% or random blood sugar >450 mg/dl
* Chronic oral steroid use
* Use of IV corticosteroid, immunosuppressive, or cytotoxic agents
* IV antibiotics
* Another ulcer within 5cm of the Index ulcer
* Cellulitis, evidence of infection, or osteomyelitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Complete closure of index wound | Up to Day 56

SECONDARY OUTCOMES:
Time to wound closure | Up to Day 56
Proportion of patients that achieve a 50% reduction or greater in wound size | Day 28
Number of product applications | Up to Day 56
Number of Adverse Events | Up to Day 56
Number of patients with worsening of wound by ≥50% increase in size | Up to Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Sharron McCulloch, Study Director — Director, Clinical Affairs
Locations (3):
- United States (3):
  - Arizona City, Arizona
  - California City, California
  - New Mexico, New Mexico

IPD SHARING:
Plan to Share IPD: No